CLINICAL TRIAL: NCT05729490
Title: Techniques and Pitfalls of Multi-Slice CT Coronary Angiography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mostafa Magdy Mahmoud, Resident of diagnostic and interventional radiology department, Sohag University Hospitals, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Soh-Med-23-01-11
Record Dates: First submitted 2023-01-18; First posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Computed Tomography Angiography; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants (Experimental)
  Interventions: Radiation: Coronary computed tomography angiography

INTERVENTIONS:
Radiation: Coronary computed tomography angiography — All patients will be subjected to:
  Two CT scans (coronary calcium scoring and angiography) using 128 or 160-row scanners with a slice thickness of 0.5 mm (Revolution Evo 128, GE Health care, Chicago, Illinois, USA) or (Aquilion 160, Canon Medical Systems, Tochigi, Japan). Calcium scoring will be performed with the use of prospective electrocardiographic gating with 400-ms gantry rotation, 120-kV tube voltage, and 300-mA tube current. For CTA, retrospective electrocardiographic gating will be used, with heart rate adjusted gantry rotations of 350 ms to 500 ms to enable adaptive multisegmented reconstruction.
  Iopromide (Ultravist 370, Bayer AG, Berlin, Germany) is the intravenous contrast medium that will be used for CTA. Beta-blockers will be given if the resting heart rate is 70 beats/min.

SUMMARY:
The goal of this study is to describe the techniques for coronary multi-slice CT angiography and to illustrate the spectrum of artifacts that can simulate coronary artery stenosis and lead to non-assessable segments using 128- and 160 multi-detector row CT scanners and discuss post-processing pitfalls with each. In addition, to review the normal anatomy and anatomic variants of the coronary arteries and discuss effective strategies for improving the diagnostic accuracy of coronary CT angiography.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients of at least 18 years of age, with suspected symptomatic CAD.

Exclusion Criteria:

* Un cooperative patients.
* Those who have allergy to iodinated contrast material or contrast-induced nephropathy,
* Elevated serum creatinine level (1.5 mg/dl) or creatinine clearance >60 ml/min.
* Atrial fibrillation.
* Aortic stenosis.
* Percutaneous coronary intervention within the past 6 months.
* Intolerance to beta-blockers.
* Body mass index > 40
* Patients with Agatston calcium scores of >400

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Number of techniques | 2 months
  The number of possible techniques used to perform CT coronary angiography
Number of pitfalls | 3 months
  The number of pitfalls that could mimic coronary artery stenosis and lead to non-assessable segments
Number of possible strategies to overcome the pitfalls of the study | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University hospitals, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maroules CD, Rajiah P, Bhasin M, Abbara S. Current Evidence in Cardiothoracic Imaging: Growing Evidence for Coronary Computed Tomography Angiography as a First-line Test in Stable Chest Pain. J Thorac Imaging. 2019 Jan;34(1):4-11. doi: 10.1097/RTI.0000000000000357. PMID 30157094
- [Background] Tridandapani S, Banait-Deshmane S, Aziz MU, Bhatti P, Singh SP. Coronary computed tomographic angiography: A review of the techniques, protocols, pitfalls, and radiation dose. J Med Imaging Radiat Sci. 2021 Nov;52(3S):S1-S11. doi: 10.1016/j.jmir.2021.08.014. Epub 2021 Sep 24. PMID 34565701
- [Background] Sun Z, Choo GH, Ng KH. Coronary CT angiography: current status and continuing challenges. Br J Radiol. 2012 May;85(1013):495-510. doi: 10.1259/bjr/15296170. Epub 2012 Jan 17. PMID 22253353
- [Background] Donnino R, Jacobs JE, Doshi JV, Hecht EM, Kim DC, Babb JS, Srichai MB. Dual-source versus single-source cardiac CT angiography: comparison of diagnostic image quality. AJR Am J Roentgenol. 2009 Apr;192(4):1051-6. doi: 10.2214/AJR.08.1198. PMID 19304713